CLINICAL TRIAL: NCT01323114
Title: The Surgical Treatment of Type 2 Diabetes Mellitus in Non-Morbidly Obese Patients: A Community Hospital Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McKenzie Health System (Other)
Responsible Party: Marcus K. Free, M.D., McKenzie Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LDE-199979-1
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; non-morbidly obese; laparoscopic duodenal exclusion
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Control Group (Active Comparator): Control group of patients who will receive conventional medical treatment for type 2 diabetes, along with regular dietary and diabetic education, under the monitoring of the study endocrinologist.
  Interventions: Other: Conventional Medical Treatment
- Surgical Treatment Group (Experimental): Experimental group in which patients will undergo the laparoscopic duodenal bypass procedure along with regular dietary and diabetic education, under the monitoring of the study endocrinologist.
  Interventions: Procedure: Laparoscopic duodenal exclusion

INTERVENTIONS:
Procedure: Laparoscopic duodenal exclusion — Laparoscopically-performed Roux-en Y intestinal bypass of the duodenum and proximal jejunum; stomach remains normal size and proximal division performed just distal to pylorus.
  Other Names: duodenal exclusion; duodenal bypass
  Arms: Surgical Treatment Group
Other: Conventional Medical Treatment — Standard of care medical treatment for type 2 diabetes to include medications and dietary management under the monitoring of the study endocrinologist.
  Other Names: control arm
  Arms: Medical Control Group

SUMMARY:
Type 2 diabetes mellitus is a chronic disease with severe long-term health consequences. In patients with type 2 diabetes mellitus who are also morbidly obese, an abundance of clinical evidence exists showing that significant clinical improvement in their diabetes occurs following certain types of bariatric, or weight loss, surgical procedures. There is additional data showing that bariatric surgical procedures that bypass the beginning of the small intestine, such as the Roux-en Y gastric bypass, can markedly improve type 2 diabetes even before significant weight loss has occurred. This early effect on type 2 diabetes prior to weight loss suggests that bypassing the beginning of the small intestine in patients who are not morbidly obese may also treat type 2 diabetes. There have been small studies outside the United States that support the concept of treating type 2 diabetes with a surgical procedure that bypasses the beginning of the small intestine without causing significant weight loss; however, data is limited in the United States and a call for comparative studies has been made internationally. The investigators propose to compare, in patients who are not morbidly obese, conventional medical treatment of type 2 diabetes to surgical treatment of type 2 diabetes using a bypass procedure that does not cause significant weight loss, the laparoscopic duodenal exclusion.

DETAILED DESCRIPTION:
Diabetes is a disease of glucose metabolism which in the United States in 2007 was estimated to effect at least 17.5 million people with type 2 diabetes mellitus accounting for approximately 90% to 95%. Poorly-controlled or treated type 2 diabetes is associated with a variety of health risks, including heart disease, stroke, renal failure, amputations,and blindness and is the seventh leading cause of death in the United States (NDIC, National Diabetes Statistics, 2011). A large number of medical treatments are available yet approximately 67% of patients in the United States with type 2 diabetes are unable to reach levels of hemoglobin A1C less than 6.5%, which is the target level set by the American Association of Clinical Endocrinologists (AACE, State of Diabetes in America, 2011). In patients with type 2 diabetes mellitus who are also morbidly obese, certain bariatric surgical procedures have shown improvement in the control of type 2 diabetes in addition to the expected weight loss effects. However, clinical investigations have pointed to a mechanism other than just weight loss in the improvement of type 2 diabetes in these patients and raised the possibility of utilizing the same mechanism in non-morbidly obese patients. Subsequent basic science research in 2004 involving a surgical bypass procedure of the proximal intestine in non-obese mice with type 2 diabetes mellitus showed remission of diabetes in the majority of mice and marked improvement over medical treatment in the remaining mice (13). Human clinical trials have been conducted in various locations worldwide and have produced similar results to the animal study; a call has been made for studies of new surgical procedures for the treatment of type 2 diabetes in IRB-approved clinical trials (39). In several studies, the duodenal exclusion, which is a procedure which bypasses the duodenum and proximal jejunum and leaves the stomach intact, has been shown to cause remission or marked improvement in type 2 diabetes mellitus without significant weight loss in non-morbidly obese patients. However, no study within the United States has compared the effect of this surgical procedure upon type 2 diabetes with the effect of conventional medical treatment of type 2 diabetes in a controlled clinical trial. In this clinical study, the investigators propose to directly compare the treatment of type 2 diabetes mellitus in non-morbidly obese humans by a surgical bypass of the duodenum and proximal jejunum to the treatment of a similar group of humans treated with conventional medical therapy. Our hypothesis is that a non-bariatric surgical procedure, the laparoscopic duodenal exclusion, will provide improved treatment of type 2 diabetes mellitus in non-morbidly obese patients when compared to conventional medical treatment. The measures of the treatment of type 2 diabetes mellitus in which a difference is expected to be observed are glycosylated hemoglobin A1C (HbA1C), fasting glucose, and insulin resistance. The investigators propose a prospective, controlled, non-randomized clinical trial to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes mellitus
* fasting blood glucose > 126 mg/dl
* on hypoglycemic medications for the treatment of type 2 diabetes
* inadequate control of diabetes with glycosylated hemoglobin A1c > 7.5
* body mass index between 20 and 35
* C-peptide level 1.0 mg/dl or higher
* ability to understand the proposed surgical treatment and its mechanism
* ability to understand the risks and benefits of the proposed surgery
* ability to commit to the study requirements for followup and education
* ability to give properly informed consent for participation

Exclusion Criteria:

* body mass index 35 or higher, or less than 20
* previous diagnosis of type 1 diabetes mellitus or mixed diabetes
* pregnancy, within one year postpartum, or currently breastfeeding
* recent (within 1 year) gastric or duodenal ulcer
* use of immunosuppressive medications or known immunosuppressive disorder
* previous gastric, duodenal, or small intestinal surgery
* inflammatory bowel disease
* treatment with anticoagulant or antiplatelet medication other than aspirin 81 mg/day
* end-stage renal disease or on dialysis
* any other serious concomitant medical condition that, in the opinion of the investigator, would compromise the safety of the patient or compromise the patient's ability to participate in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | One year
  The primary outcome is the difference in hemoglobin A1C between the surgical treatment arm and the conventional medical treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus K. Free, M.D., Principal Investigator — McKenzie Health System; Steve Barnett, M.S., Study Director — McKenzie Health System
Locations (1):
- McKenzie Health System, Sandusky, Michigan, United States